CLINICAL TRIAL: NCT00169832
Title: A Multicenter Randomized Double-Blind Trial Comparing Rosiglitazone to Placebo for the Prevention of Atherosclerosis Progression After Coronary Bypass Surgery in Diabetic Patients
Brief Title: Vein-Coronary Atherosclerosis And Rosiglitazone After Bypass Surgery: The VICTORY Trial
Acronym: VICTORY
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Laval University (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Olivier F Bertrand, MD PhD, Hopital Laval
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 49653/416; ISRCTN54136716
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2008-10-10 (Estimated); Status verified 2008-10

CONDITIONS: Diabetes; Coronary Artery Bypass Grafting
Keywords: Atherosclerosis progression; Ischemic heart disease; Saphenous vein graft; Metabolic risk factors; Rosiglitazone
MeSH Terms: conditions — Diabetes Mellitus; Myocardial Ischemia | interventions — Rosiglitazone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rosiglitazone (Avandia) (Experimental)
  Interventions: Drug: Rosiglitazone or placebo
- Placebo (Placebo Comparator)
  Interventions: Drug: Rosiglitazone or placebo

INTERVENTIONS:
Drug: Rosiglitazone or placebo — Rosiglitazone 4 to 8 mg/day or placebo, for 12 months
  Other Names: Avandia

SUMMARY:
HYPOTHESES

* Rosiglitazone in diabetic patients with previous coronary bypass surgery may prevent or slow the progression of atherosclerosis in SVGs and native coronary arteries.
* Rosiglitazone has favorable effects on adipose tissue distribution variables as well as on thrombosis, pro-inflammatory, and lipid profiles in diabetic patients after coronary bypass artery surgery.
* Rosiglitazone therapy influences favorably metabolism and clinical outcomes in diabetic patients after coronary artery bypass surgery.

OBJECTIVES

* PRIMARY To assess the efficacy of rosiglitazone to reduce atherosclerosis progression in vein grafts in diabetic patients after coronary bypass surgery by using IVUS imaging after a 12 mo follow-up.
* SECONDARY

  * To prospectively compare the secondary IVUS endpoints.
  * To prospectively compare the angiographic endpoints.
  * To prospectively compare the metabolic risk factor endpoints.
  * To prospectively compare the body composition and distribution endpoints.
  * To prospectively compare the clinical outcomes of rosiglitazone versus standard care using composite endpoints.

DETAILED DESCRIPTION:
STUDY DESIGN

This is a prospective multicenter randomized placebo-controlled double-blind trial assessing the efficacy and safety of rosiglitazone in the prevention of atherosclerosis progression in vein grafts and native coronary arteries of diabetic patients. Stable diabetic patients with previous coronary bypass surgery (≥ 1 year ≤ 10 years) will be screened. After baseline evaluation, all eligible patients will undergo baseline coronary angiogram. IVUS will be performed in a segment length of at least 40 mm in a SVG suitable for IVUS analysis and in a segment length of at least 20 mm in the anastomosed native coronary artery corresponding to the SVG chosen. Following the IVUS procedure, patients will be randomized to either rosiglitazone treatment or to placebo in addition to their standard clinical care. Study drug will be titrated over an 8-week period up to a dose of 8 mg/day (or to maximum tolerated dose). The patients will receive the study drug or the placebo for 50-54 weeks in a double-blind manner. At the beginning and at 2, 4, 6, 8, 10 and 12 months of treatment, patients will be subjected to a set of morphological, physiological and metabolic evaluations. At the final visit (12 months), patients will also be submitted to IVUS and angiography.

ELIGIBILITY:
Inclusion Criteria:

AT SCREENING:

1. Male or female, aged ≥ 40 years & ≤ 75 years.
2. Women of childbearing potential with contraceptive measure, or of non-childbearing potential or surgically sterile.
3. Type 2 diabetes mellitus.
4. Patients with no new medication for hyperglycemia and no change in dose of oral hypoglycemic medication within the last 3 mo prior to screening.
5. Diabetic patients with ischemic heart disease and CABG with at least one SVG (≥1 yr & ≤10 yrs).
6. Patient agrees to participate.
7. Patient legally capable of giving consent and understand what participation in study entails, potential risks and benefits, freedom to withdraw without any prejudice to subsequent medical arrangement or treatment, sign an ICF prior to any protocol specific procedure.

AT IVUS & ANGIOGRAPHY (VISIT 2):

Subject eligible if at least 1), 2) and 3) of the following criteria apply:

1. Patient with at least 1 patent SVG.
2. Segment length of at least 40 mm in SVG suitable for IVUS.
3. Reference of target (SVG) diameter ≥ 2.5 mm.

   If anastomosed native coronary artery or non grafted coronary artery can be evaluated, the following criteria must be met:
4. Reference of target anastomosed native coronary artery or non grafted coronary artery diameter≥ 2.5 mm.
5. Segment length of at least 20 mm in anastomosed native coronary artery corresponding to SVG chosen or, in case of impossibility of performing IVUS in the anastomosed coronary artery, a non grafted coronary artery (≥ 30 mm length segment) might be used for reference.

Exclusion Criteria:

AT SCREENING:

1. Clinically significant abnormality at screening tests & exams.
2. Type 1 diabetes or history of diabetic ketoacidosis.
3. Uncontrolled type 2 diabetes mellitus.
4. Recent MI or ACS (≤ 90 days).
5. History of hypersensitivity to thiazolidinediones (TZD) or compounds of similar chemical structures.
6. Last LVEF≤ 35%.
7. SBP>170mmHg or DBP>100mmHg at screening/baseline should be appropriately treated and under control prior to randomization.
8. Unstable or Canadian Cardiovascular Society class III and IV angina, acute heart failure or congestive heart failure (NYHA class III and IV).
9. History of hepatocellular reaction/severe oedema/other potentially fluid-related AE associated with use of any TZD or PPAR-γ agonist.
10. Hepatic disease.
11. Renal dysfunction.
12. Anemia.
13. TG ≥ 10 mmol/L.
14. History of PCI in all SVG(s).
15. Known occlusion(s) of all SVG(s).
16. Treatment involving TZD within 3 mo prior to screening.
17. Chronic use (≥ 6 mo) of insulin for glycemic control at any time in the past or administration of insulin any time within the last 12 mo.
18. Allergy to contrast agents.
19. Current intake of anorectic agents or have been taken off an anorectic agent or equivalent within 3 mo prior to screening.
20. Patients for whom oral or injectable corticosteroids are used on a regular or recurrent basis.
21. Recent history/suspicion of current drug abuse or alcohol abuse within last 6 mo.
22. Women breast feeding, pregnant, or planning to become pregnant during conduct of trial and for 30 days after study completion.
23. Other illness that precludes survival.
24. History of malignancy within the last 5 yrs.
25. Concurrent participation in other investigational device or drug studies and/or having received any experimental therapeutic agents within 30 days of the screening.
26. Use of any investigational drug for glycemic control within 3 mo of the screening.
27. Patient travelling out of town/country for periods exceeding 2 mo.
28. Medical condition which may interfere with intake and/or absorption of study medication.
29. Patients unwilling or unable to comply with procedures.
30. Recent major surgery within 90 days of the screening.

AT IVUS AND ANGIOGRAPHY (VISIT 2):

1. PCI was performed on the target segment(s) after CABG.
2. Target SVG and/or target native coronary artery show ≥ 50% angiographic lesion precluding IVUS.
3. Thrombus/thrombus aspect in target vessels.
4. Target vessel has been subjected to surgical endarterectomy.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 193 (Actual)
Dates: Start 2003-06; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Change in plaque volume in one SVG (by IVUS) | 12 months

SECONDARY OUTCOMES:
1 Change in plaque volume in segment of anastomosed coronary artery | 12 months
2 Changes in lumen and total vessel volumes and lumen plaque total vessel areas in SVG and coronary segments | 12 months
3 Changes in qualitative plaque characterization in the SVG and coronary segments | 12 months
4 Patients showing atherosclerosis changes | 12 months
5 Atherosclerosis changes concordance and discordance | 12 months
6 New occlusions in native coronary arteries or SVGs | 12 months
7 Changes in reference and minimum lumen diameters of the SVG | 12 months
8 Per patient percentage of initially patent SVGs that had significant progression of atherosclerosis at the site of greatest change at follow-up | 12 months
9 Changes of indices for comprehensive lipid thrombosis and pro-inflammatory profiles as well as glucose-insulin homeostasis, microalbuminuria, adhesion molecules, adipokines, and other markers relevant to the evaluation and management of cardiovascular | 12 months
10 Changes in abdominal areas and volumes of adipose tissue areas | 12 months
11 Changes in body composition, body weight, waist circumference and BMI | 12 months
12 Clinical laboratory parameters, physical examinations, vital signs, ECGs, concomitant medication and adverse events | 12 months
13 Death, MI, TIA, stroke, hospitalization and ischemia-driven interventions | 12 months
14 Fluid retention | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Olivier F Bertrand, MD, PhD, Principal Investigator — Laval Hospital Research Center; Jean-Pierre Despres, PhD, Principal Investigator — Laval Hospital Research Center; Paul Poirier, MD, PhD, Principal Investigator — Laval Hospital Research Center
Locations (9):
- Canada (6):
  - QEII Health Sciences Center - Halifax Infirmary, Halifax, Nova Scotia
  - Hamilton Health Sciences - Mc Master Clinic, Hamilton, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - CRMSBC, Bonaventure, Quebec
  - CHUM Notre-Dame Hospital, Montreal, Quebec
  - Laval Hospital, Sainte-Foy, Quebec
- Spain (3):
  - Hospital Del Mar, Barcelona
  - Hospital Universitari Vall D'Hebron, Barcelona
  - Hospital Universitarion Son Dureta, Palma de Mallorca

REFERENCES:
- [Derived] Bertrand OF, Poirier P, Rodes-Cabau J, Rinfret S, Title LM, Dzavik V, Natarajan M, Angel J, Batalla N, Almeras N, Costerousse O, De Larochelliere R, Roy L, Despres JP; VICTORY Trial Investigators. Cardiometabolic effects of rosiglitazone in patients with type 2 diabetes and coronary artery bypass grafts: A randomized placebo-controlled clinical trial. Atherosclerosis. 2010 Aug;211(2):565-73. doi: 10.1016/j.atherosclerosis.2010.06.005. Epub 2010 Jun 11. PMID 20594555